CLINICAL TRIAL: NCT06943417
Title: Safety and Efficacy of Endoscopic Full Thickness Biopsy With Over the Scope Clip in Patients With Chronic Intestinal Pseudo-obstruction: A Single-Center, Single-Arm, Open-label, Interventional Trial
Brief Title: Safety and Efficacy of Endoscopic Full Thickness Biopsy in Patients With Chronic Intestinal Pseudo-obstruction
Acronym: EFTB-CIPO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International University of Health and Welfare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-CN-021; UMIN000057266 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2025-03-13; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Chronic Intestinal Pseudo-obstruction
Keywords: Chronic intestinal pseudo-obstruction; Endoscopic full thickness biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Over the scope clip (Experimental)
  Interventions: Device: Over the scope clip

INTERVENTIONS:
Device: Over the scope clip — over the scope clip group

SUMMARY:
To evaluate the safety and efficacy of endoscopic full thickness biopsy for the diagnostic purpose of chronic intestinal pseudo-obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pseudo intestinal obstruction or suspected chronic pseudo intestinal obstruction
* Patients who are 18 years of age or older at the time of obtaining consent
* Gender: Any

Exclusion Criteria:

* Patients for whom it is difficult to perform endoscopy
* Patients who cannot obtain consent
* Patients with serious renal, hepatic, or cardiac disease
* Patients who are participating in other clinical research, except for observational research.
* Other patients whom the principal investigator or subinvestigator determines to be inappropriate to conduct this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of total perforations (intraoperative and delayed perforations) | Immediately after the intervention
  Percentage of total perforations (intraoperative and delayed perforations)

SECONDARY OUTCOMES:
Intraoperative perforation rate | Under procedure
  Intraoperative perforation rate
Rate of delayed perforation | Periprocedural
  Rate of delayed perforation
Intraoperative complications | Under procedure
  Intraoperative complications
Intraoperative death rate | Under procedure
  Intraoperative death rate
Examination time | Under procedure
  Examination time
Macroscopic specimen size | Immediately after procedure
  Macroscopic specimen size
Findings of tissue specimens | Immediately after procedure
  Findings of tissue specimens
Whether tissue evaluation is acceptable for biopsy purposes | Immediately after procedure
  Whether tissue evaluation is acceptable for biopsy purposes
Ratio of postoperative complications | Immediately after procedure
  Ratio of postoperative complications
Time or days of fluid intake postoperatively | From date of procedure until the date of first fluid intake assessed up to 12 months
  Time or days of fluid intake postoperatively
Time or number of days of food intake after procedure | From date of procedure until the date of first food intake assessed up to 12 months
  Time or number of days of food intake after procedure
Length of hospital stay | From date of procedure until the date of discharge assessed up to 12 months
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Takaomi Kessoku, M.D., Ph.D., Principal Investigator — International university of health and welfare Narita hospital
Locations (1):
- International university health and welfare Narita hospital, Narita, Japan

IPD SHARING:
Plan to Share IPD: No